CLINICAL TRIAL: NCT02658084
Title: A Phase I/II Study to Evaluate the Safety and Efficacy of Vinorelbine With Trastuzumab Emtansine in Pre-Treated HER2-Positive Metastatic Breast Cancer
Brief Title: Vinorelbine With Trastuzumab Emtansine in Pre-Treated HER2-Positive Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to low accrual and toxicity concerns.
Sponsor: University of Miami (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Reshma Mahtani, Assistant Professor of Clinical, University of Miami
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20151055
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
Keywords: HER2-Positive; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: T-DM1 + Vinorelbine (Experimental): One cycle of Trastuzumab Emtansine (T-DM1)/Vinorelbine combination treatment is defined as 21-days (i.e. 3 weeks). The recommended (starting) dose of trastuzumab emtansine is 3.6 mg/kg given as an intravenous infusion on Day 1 of every 21-day cycle. The starting dose of Vinorelbine is 22.5 mg/m2 given as a direct intravenous push over 6-10 minutes on day 1 and day 8 of every 3-week (i.e. 21-day) cycle. Participants will be treated until documented disease progression or other criteria for discontinuation. Approximately 15 to 21 patients will be needed to establish the recommended phase II dose (RP2D).
  Interventions: Drug: Vinorelbine; Drug: Trastuzumab Emtansine
- Phase 2: T-DM1 + RP2D Vinorelbine (Experimental): One cycle of trastuzumab emtansine (T-DM1)/vinorelbine combination treatment is defined as 21-days (i.e. 3 weeks). Participants will receive the recommended Phase 2 Dose (RPSD) of Vinorelbine with the fixed dose (3.6 mg/kg) of Trastuzumab Emtansine. Participants will be treated until documented disease progression or other criteria for discontinuation. Up to 35 patients will be treated at the RP2D (MTD) including 6 patients treated at RP2D in phase I.
  Interventions: Drug: Vinorelbine; Drug: Trastuzumab Emtansine

INTERVENTIONS:
Drug: Vinorelbine — Administered as an intravenous infusion on Day 1 and Day 8 of every 21-day cycle.
  Other Names: Vinorelbine tartrate; Navelbine
Drug: Trastuzumab Emtansine — Administered as an intravenous infusion on Day 1 of every 21-day cycle.
  Other Names: Kadcyla; T-DM1; Trastuzumab-MCC-DM1

SUMMARY:
The study proposes to evaluate the safety and efficacy of the combination of trastuzumab emtansine (T-DM1) and vinorelbine in HER2+ metastatic breast cancer patients.

DETAILED DESCRIPTION:
This is a Phase I/II, single arm, open-label clinical trial designed to establish the recommended phase II dose (RP2D) of vinorelbine with a fixed dose of trastuzumab emtansine. The study will also evaluate the safety and efficacy of the RP2D in patients with human epidermal growth factor receptor 2 (HER2)-positive metastatic, locally advanced, or unresectable breast cancer. The study will be opened to accrual at the University of Miami Sylvester Comprehensive Cancer Center (SCCC) main campus and constituent satellite sites, Deerfield Beach and Plantation.

This phase I/II study will have a total of 50 enrolled patients, taking into account 10% drop-out in the phase II follow-up. The duration anticipated to enroll all study subjects in Phase I/II is 2 years. The estimated duration for the Investigators to complete this study (Phase I/II) is 4.5 to 5 years.

For the phase I portion, standard 3+3 dose escalation/de-escalation design will be applied. Approximately 15 to 21 patients will be needed to establish the recommended phase II dose (RP2D). For the phase II portion of the study, up to 35 patients will be treated at the RP2D (MTD) including 6 patients treated at RP2D in phase I. Patients may remain on treatment with the combination until disease progression or unmanageable toxicity.

Tumor assessments will be conducted every 6 weeks (±7 days) to week 18. Thereafter, these assessments will be done every 12 weeks (±7 days). These will shall occur regardless of dose delays or dose interruptions, until Investigator-assessed progressive disease (PD), or death, whichever occurs first. More frequent tumor assessments may be performed as clinically indicated, at the discretion of the treating Investigator.

For the phase II portion of the study - patients who discontinue treatment for reasons other than PD will continue to have required tumor assessments completed until PD or the initiation of a new therapy. Once patients have progressed, they will be followed for survival approximately every 3 months for at least 3 years. Subsequent anti-cancer therapies will be documented until study completion.

Patients who are discontinued from study treatment will return for the Study Treatment Discontinuation Visit approximately 30 days (±7 days) after the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented breast cancer.
2. Metastatic or unresectable locally advanced/recurrent breast cancer.
3. HER2-positive disease documented as: Immunohistochemistry (IHC) 3+ positive, and/or Fluorescence in situ hybridization (FISH) ≥ 2.0, and/or gene copy number greater than 6, on previously collected tumor or metastatic site. IHC testing, FISH assay(s), and gene copy number may all have been performed; however, a positive result from only one of the above is required for eligibility.
4. Documented disease progression on the last regimen by radiographic measurement (progression demonstrated by tumor markers only is unacceptable).
5. Documented disease progression (by investigator assessment) after at least one regimen of HER2-directed therapy in the metastatic or unresectable locally advanced/recurrent setting.
6. For patients with hormone receptor-positive disease: disease progression or recurrence in any setting on prior hormonal therapy, given with or without HER2 directed therapy.
7. Measurable or bone only disease.
8. Prior treatment with a taxane, in the neoadjuvant, adjuvant, locally advanced or metastatic setting.
9. A minimum of 6 weeks of prior trastuzumab for the treatment of metastatic or unresectable locally advanced/recurrent disease is required.
10. Prior use of Pertuzumab in any setting is permitted (but not required).
11. Prior use of Lapatinib in any setting is permitted (but not required).
12. Age ≥ 18 years
13. Life expectancy ≥ 3 months
14. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. See Appendix C for details.
15. Patients must have normal organ and marrow function as defined below:

    * absolute neutrophil count (ANC) >1,500 cells/mm3
    * platelets >100,000 cells/mm3
    * hemoglobin > 9.0 g/dL (Patients are permitted to receive transfused red blood cells to achieve this level.)
    * total bilirubin ≤1.5 X institutional upper limit of normal (ULN) [Note: For patients with previously documented Gilbert's syndrome, total bilirubin ≤ 3 mg/dL.]
    * Aspartate aminotransferase (AST/SGOT) ≤ 2.5 X ULN
    * Alanine aminotransferase (ALT/SGPT) ≤ 2.5 X ULN
    * alkaline phosphatase (alk phos) ≤ 2.5 X ULN
    * serum creatinine < 1.5 X ULN
16. International normalized ratio (INR) < 1.5 X ULN
17. Left ventricular ejection fraction (LVEF) ≥ 50% by either echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA).
18. Negative results of serum pregnancy test for premenopausal women of reproductive capacity and for women < 12 months after menopause. For men and women of childbearing potential, agreement by the patient and/or partner to use two effective non-hormonal forms of barrier contraception at the same time, throughout treatment on study. Women should agree to continued use for at least 90 days after the end of treatment. Men should agree to continued use for at least 7 months after the end of treatment. Examples of non-hormonal barrier contraception include: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicide.
19. Ability to understand and willingness to sign a written informed consent and HIPAA document.

Exclusion Criteria:

1. Chemotherapy ≤21 days prior to first dose of study treatment
2. If last dose of trastuzumab was:

   * 6mg/kg then ≤21 days prior to first dose of study treatment
   * 4mg/kg then ≤14 days prior to first dose of study treatment
   * 2mg/kg then ≤7 days prior to first dose of study treatment
3. Lapatinib ≤14 days prior to first dose of study treatment
4. Pertuzumab ≤21 days prior to first dose of study treatment
5. Hormone therapy ≤7 days prior to first dose of study treatment
6. Investigational therapy or any other such experimental therapy ≤28 days prior to first dose of study treatment
7. Prior treatment with trastuzumab emtansine, (on or off a study protocol)
8. Prior use of vinorelbine (in any setting).
9. Previous radiotherapy for the treatment of unresectable, locally advanced, recurrent or metastatic breast cancer is not allowed if:

   * The last fraction of radiotherapy has been administered within 14 days prior to study enrollment
   * More than 25% of marrow-bearing bone has been irradiated
10. Brain metastases that are untreated or symptomatic, or require any radiation, surgery, or continued steroid therapy to control symptoms from brain metastases within 14 days of study enrollment.
11. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins.
12. History of exposure to the following cumulative doses of anthracyclines:

    * Doxorubicin ≥550mg/m2
    * Liposomal doxorubicin >500 mg/m2
    * Epirubicin >900 mg/m2
    * Mitoxantrone > 120 mg/m2
    * If another anthracycline, or more than one anthracycline, has been used, the cumulative dose must not exceed the equivalent of ≥550 mg/m2 doxorubicin.
13. Current peripheral neuropathy of Grade ≥3 per the NCI CTCAE, v4.0
14. The patient has not recovered from any other acute toxicity (to Grade ≤1 as per NCI CTCAE v4.03) prior to study enrollment.
15. History of other malignancy within the last 3 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome.
16. Cardiopulmonary Function Criteria:

    * Current unstable ventricular arrhythmia requiring treatment
    * History of symptomatic congestive heart failure (CHF) as per New York Heart Association (NYHA) Classes II-IV; see Appendix D for details.
    * History of myocardial infarction or unstable angina within 6 months of study enrollment
    * History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment
    * Severe dyspnea at rest due to complications of advanced malignancy or requiring current continuous oxygen therapy
17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)

    * Major surgical procedure or significant traumatic injury within 28 days -before enrollment or anticipation of the need for major surgery during the course of study treatment
    * Current pregnancy or lactation
    * Current known uncontrolled active infection with HIV, hepatitis B, and/or hepatitis C virus
18. Any uncontrolled, intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.
19. Any other serious medical or psychiatric illness/condition likely in the judgment of the Investigator(s) to interfere or limit compliance with study requirements/treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Mahtani, DO, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase 1: T-DM1 + Vinorelbine | Phase 2: T-DM1 + RP2D Vinorelbine
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Study Termination | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only Phase 1 enrolled participants, however, the study was terminated early. The Phase 2 arm did not open to accrual.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: T-DM1 + Vinorelbine | Phase 2: T-DM1 + RP2D Vinorelbine | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 - Maximum Tolerated Dose (MTD) of Vinorelbine in Combination With a Fixed Dose of Trastuzumab Emtansine.
Description: Identifying the Maximum Tolerated Dose (MTD) of Vinorelbine combined with a fixed dose of Trastuzumab Emtansine to be recommended for the phase II portion of the study (RP2D).
Time Frame: 2 years
Population: Approximately 15 to 21 participants would be needed to establish the recommended phase II dose (RP2D). Only 2 participants were enrolled therefore the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) were not determined.
Arm/Group | Phase 1: T-DM1 + Vinorelbine
Number analyzed (Participants) | 0

2. Primary Outcome: Phase 2 - Rate of Progression-Free Survival (PFS)
Description: Rate of Progression-Free Survival (PFS) in participants receiving the RP2D of vinorelbine in combination with Trastuzumab Emtansine therapy. PFS is defined as the time from date from first treatment received on study until documented disease progression or death (by any cause, in the absence of progression). In progression-free patients, PFS will be censored at the last evaluable tumor assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
Time Frame: Up to 5 years
Population: The Phase 2 arm did not open to accrual. No participants were enrolled to Phase 2.
Arm/Group | Phase 2: T-DM1 + RP2D Vinorelbine
Number analyzed (Participants) | 0

3. Primary Outcome: Phase 1 - Rate of Participants Experiencing Adverse Events
Description: Rate of participants experiencing adverse events including dose-limiting toxicities (DLTs) and serious adverse events (SAEs).
Time Frame: 18 months
Population: For adverse events, participants who received at least one dose of study therapy. For dose-limiting toxicities, participants who experienced a dose-limiting toxicity during the first two cycles of study therapy.
Measure: Number; unit: participants
Arm/Group | Phase 1: T-DM1 + Vinorelbine
Number analyzed (Participants) | 2
participants
  Dose-limiting toxicities (DLTs) | 2
  Adverse events (AEs) | 2

4. Secondary Outcome: Phase 2 - Clinical Benefit Rate (CBR)
Description: Rate of participants achieving best overall response of complete response (CR), partial response (PR) or stable disease (SD) for >/= 6 months on protocol therapy, according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria
Time Frame: Up to 5 years
Population: The Phase 2 arm did not open to accrual. No participants were enrolled to Phase 2.
Arm/Group | Phase 2: T-DM1 + RP2D Vinorelbine
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase 2 - Overall Survival (OS) Rate
Description: Overall Survival (OS) is defined as the elapsed time from date from first treatment received on study to death or date of censoring. Patients alive or those lost to follow-up will be censored at the last date of contact (or last date known to be alive).
Time Frame: Up to 5 Years
Population: The Phase 2 arm did not open to accrual. No participants were enrolled to Phase 2.
Arm/Group | Phase 2: T-DM1 + RP2D Vinorelbine
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase 2 - Objective Response Rate (ORR)
Description: Rate of participants achieving a best overall response of complete response (CR) or partial response (PR) to protocol therapy according to Response Evaluation Criteria in Solid Tumors (RECIST) v. 1.1 criteria.
Time Frame: Up to 5 Years
Population: The Phase 2 arm did not open to accrual. No participants were enrolled to Phase 2.
Arm/Group | Phase 2: T-DM1 + RP2D Vinorelbine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Phase 1: T-DM1 + Vinorelbine
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: T-DM1 + Vinorelbine (N=2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: T-DM1 + Vinorelbine (N=2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypercapnia (Blood and lymphatic system disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (6)
Fever (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Platelet count decreased (Investigations) | 2 (3)
Somnolence (Nervous system disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hypochloremia (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early study termination by mutual decision of the Sponsor and the Investigator due to lower than expected accrual and toxicities concerns. Only the Phase 1 arm opened to accrual; Phase 2 did not open to accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT02658084/Prot_SAP_000.pdf